CLINICAL TRIAL: NCT02358850
Title: Post-tonsillectomy Pain Control in Adults: a Randomized Prospective Study
Brief Title: Post-tonsillectomy Pain Control in Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0658-14-FB
Record Dates: First submitted 2015-01-14; First posted 2015-02-09 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Hemorrhage; Body Weight Changes
Keywords: Tonsillectomy; Adenoidectomy
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Hemorrhage; Body Weight Changes | interventions — oxycodone-acetaminophen; Hydrocodone; Acetaminophen; Oxycodone; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tonsillectomy and Norco (Active Comparator): This represents patients who will be randomized (1:3 chance) to postoperative pain control with Norco (Hydrocodone and Acetaminophen)
  Interventions: Drug: Norco (Hydrocodone and Acetaminophen)
- Tonsillectomy and Percocet (Active Comparator): This represents patients who will be randomized (1:3 chance) to postoperative pain control with Percocet (Oxycodone and Acetaminophen)
  Interventions: Drug: Percocet (Oxycodone and Acetaminophen)
- Tonsillectomy and Dilaudid + Tylenol (Active Comparator): This represents patients who will be randomized (1:3 chance) to postoperative pain control with Dilaudid (hydromorphone) and Tylenol (Acetaminophen)
  Interventions: Drug: Dilaudid (hydromorphone); Drug: Tylenol (Acetaminophen)

INTERVENTIONS:
Drug: Norco (Hydrocodone and Acetaminophen) — Norco (Hydrocodone and Acetaminophen) 5/325 mg tab Take 1-2 tabs by mouth every 4-6 hours PRN (as needed) pain following Tonsillectomy for 14 days
  Other Names: Norco
  Arms: Tonsillectomy and Norco
Drug: Percocet (Oxycodone and Acetaminophen) — Percocet (Oxycodone and Acetaminophen) 5/325 mg tab Take 1-2 tabs by mouth every 4-6 hours PRN pain following Tonsillectomy for 14 days
  Other Names: Percocet
  Arms: Tonsillectomy and Percocet
Drug: Dilaudid (hydromorphone) — Dilaudid (hydromorphone) 2 mg tab Take 1-2 tabs by mouth every 4-6 hours PRN pain following Tonsillectomy for 14 days
  Other Names: Dilaudid
  Arms: Tonsillectomy and Dilaudid + Tylenol
Drug: Tylenol (Acetaminophen) — Tylenol (Acetaminophen) 325 mg tab Take 1-2 tabs by mouth every 4-6 hours PRN pain following Tonsillectomy for 14 days
  Other Names: Tylenol
  Arms: Tonsillectomy and Dilaudid + Tylenol

SUMMARY:
This is a randomized prospective study to determine the optimal postoperative pain medication regimen for adults (18 years old and older) undergoing tonsillectomy with or without adenoidectomy for chronic tonsillitis and/or snoring and/or obstructive sleep apnea. All participants will undergo the same tonsillectomy surgical technique (with or without adenoidectomy) under general anesthesia and be randomized to one of three postoperative pain control regimens (all of which are commonly used pain medications for post-tonsillectomy pain):

1. Norco (Hydrocodone and Acetaminophen)
2. Percocet (Oxycodone and Acetaminophen)
3. Dilaudid and Tylenol (Acetaminophen)

Participants will be discharged home the day of surgery and will be sent home with questionnaires to assess their daily pain level, oral intake, amount of nausea/vomiting, and amount of pain medications taken for the 14 days following their surgery. Data will be collected and analyzed to determine if there is a difference in pain levels or oral intake or nausea/vomiting in the different pain regimen groups. Secondary endpoints will include weight change from preoperative weight to weight at 2-3 weeks after surgery in addition to postoperative complications including visits to the Emergency Department and post-tonsillectomy bleed rates.

Participants will be seen 1-2 weeks following their surgery in the ENT (Ear, Nose and Throat) clinic per normal postoperative protocol and will not require any specific clinic visits related to this study.

DETAILED DESCRIPTION:
Hypotheses

* There is an optimal pain control regimen for post-tonsillectomy pain control in adults
* Post-tonsillectomy pain levels in adults peak around postoperative day number seven
* Post-tonsillectomy adults return very slowly to normal (pre-surgery) oral intake and diet

Purpose

* To assess daily post-tonsillectomy pain level in adults for the two weeks after surgery
* To determine if there is an optimal post-tonsillectomy pain control regimen in adults for the two weeks after surgery
* To determine oral intake levels in post-tonsillectomy adults for the two weeks after surgery
* To determine daily amounts of nausea/vomiting in post-tonsillectomy adults for the two weeks after surgery
* To determine the change in weight in the two to three weeks after surgery

Study Background Tonsillectomy (with or without adenoidectomy) is a very common procedure in children and adults. The most common indications for tonsillectomies include chronic tonsillitis and/or obstructive sleep apnea. While many studies have examined the optimal postoperative pain control regimen in children, the optimal pain control regimen in adults remains poorly studied and understood.

Literature regarding post-tonsillectomy pain in adults has primarily focused on the specific tonsillectomy surgical technique (there are many) rather than the exact medications used for pain control. Interestingly, some of these aforementioned studies did not include the name, type or quantity of pain medications given to their patients when the primary study endpoint was pain. Additional studies have examined the role of steroids, antibiotics, and/or pain medications given by Anesthesia while a patient is anesthetized and undergoing tonsillectomy to determine if this can reduce postoperative pain. IV steroids given perioperatively to adults undergoing tonsillectomy have less pain, nausea, and vomiting in the first few days after tonsillectomy. IV steroids are now routinely given before tonsillectomy by most practicing Otolaryngologists, including our senior authors.

There are a limited number of studies looking at actual postoperative pain control regimens in adults. Most of these studies are limited in that they only looked at the first 24 hours following surgery rather than trending pain levels for the first week or two after surgery. Additional studies are limited because they are observational or prospective without comparative pain regimen groups (i.e. they gave all patients the same medications asked them their daily pain levels).

Furthermore, a majority of studies involving postoperative pain control used a "cold steel" technique tonsillectomy, which is uncommonly practiced in the United States by Otolaryngologists, who prefer the use of electrocautery devices for tonsillectomy. It is well known and accepted that cautery causes more postoperative pain due to thermal tissue injury, however it allows for a straightforward surgery with better intraoperative control of bleeding. Furthermore, randomized prospective studies for postoperative pain control following cautery tonsillectomy are lacking in the literature.

It is well known that the expected recovery period for adults is 2-4 weeks, during which they cannot work or do any strenuous activity. We would argue that the first 24 hours after tonsillectomy is actually better tolerated by adults because they have received high potency narcotics (usually through their IV) during and right after surgery. Therefore a more meaningful time period to study would be postoperative day number 1 - 14, when the patient is at home and the pain is most severe (most patients state that their pain peaks around postoperative number 5-7). Pain control is incredibly important issue in the post-tonsillectomy patient. If they have too much pain, they will not drink or eat enough to stay hydrated and nourished. This can lead to electrolyte abnormalities and dehydration requiring visits to the Emergency Department with or without admission to the hospital.

The purpose of this study is to evaluate post-tonsillectomy pain control in adults using three randomized medication regimens. All patients would undergo the same surgical technique to avoid confounding variables. Surgeries would be performed by Otolaryngology - Head and Neck Surgery Residents under the direct supervision of Otolaryngology staff attending surgeons. All of the proposed pain regimens are commonly accepted regimens used by practicing Otolaryngologists for adults.

Patients would be asked to complete a questionnaire that numerically evaluates their daily: pain level, amount of oral intake, amount of nausea/vomiting, and amount of pain medications used. They would asked to mail in their results or return the clinic. Additional information would be collected from the patients and/or their medical records including visits to the emergency department, readmissions to the hospital, and postoperative complications including post-tonsillectomy bleeding. Data would be compiled and analyzed to determine the typical postoperative pain levels, daily oral intake level, and to compare the different pain regimens to determine if one is superior.

It is important to note that there are accepted risks of general anesthesia and undergoing tonsillectomy with or without adenoidectomy. Participation in this study would not change any of the accepted risk of undergoing the surgical procedure. The risks commonly discussed with patients before tonsillectomy with or without adenoidectomy include failure to resolve chronic throat infections, failure to resolve obstructive sleep apnea, voice changes after surgery, damage to lips/teeth/tongue, taste changes, dehydration, need to return to the emergency department, need for admission to the hospital, and 3-5% risk of post-tonsillectomy bleeding that may result in need for additional surgical procedures and/or blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Surgical indications: Chronic tonsillitis, Snoring, Sleep apnea
* Surgical procedure: Tonsillectomy with monopolar cautery, hemostasis with monopolar cautery and/or suction cautery. The surgical procedure can also include Adenoidectomy with suction cautery

Exclusion Criteria:

* Additional surgical procedures (i.e. UPPP (uvulopalatopharyngoplasty), septoplasty, inferior turbinate reduction) during same surgery
* Pregnant females
* Indications: Suspected malignancy
* History of chronic pain or daily pain medication used for another medical problem
* History of liver disease
* Contraindications to preoperative Decadron
* Contraindications to pain regimen medications (Tylenol, Norco, Percocet, Dilaudid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Daily pain level | Postoperative day 1
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 2
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 3
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 4
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 5
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 6
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 7
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 8
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 9
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 10
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 11
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 12
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 13
  Daily pain level on scale from 0-10
Daily pain level | Postoperative day 14
  Daily pain level on scale from 0-10

SECONDARY OUTCOMES:
Daily oral liquid intake | Postoperative day 1
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 2
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 3
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 4
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 5
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 6
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 7
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 8
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 9
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 10
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 11
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 12
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 13
  Daily estimation of cups of liquids consumed
Daily oral liquid intake | Postoperative day 14
  Daily estimation of cups of liquids consumed
Daily nausea/vomiting | Postoperative day 1
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 2
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 3
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 4
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 5
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 6
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 7
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 8
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 9
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 10
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 11
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 12
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 13
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Daily nausea/vomiting | Postoperative day 14
  Daily amount of nausea/vomiting with a scale from 0 - 4. 0 = no nausea
  1. = mild nausea
  2. = significant nausea and/or dry heaving
  3. = vomiting
Weight Change from Baseline | Preoperative weight compared to postoperative weight at 2-3 weeks after surgery
  Weight change comparing preoperative weight (kg) to postoperative weight (kg) at 2-3 weeks after surgery
Visit to emergency department after surgery | Within 14 days after surgery
  Yes/No answer for if patient needed to visit the emergency department after surgery for any reason related to their surgery
Post tonsillectomy hemorrhage | Within 14 days after surgery
  If patient had a post tonsillectomy hemorrhage and if any treatment was needed

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Pate, M.D., Principal Investigator — University of Nebraska Medical Center Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- University Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Lee SW, Jeon SS, Lee JD, Lee JY, Kim SC, Koh YW. A comparison of postoperative pain and complications in tonsillectomy using BiClamp forceps and electrocautery tonsillectomy. Otolaryngol Head Neck Surg. 2008 Aug;139(2):228-34. doi: 10.1016/j.otohns.2008.04.004. PMID 18656720
- [Background] Parsons SP, Cordes SR, Comer B. Comparison of posttonsillectomy pain using the ultrasonic scalpel, coblator, and electrocautery. Otolaryngol Head Neck Surg. 2006 Jan;134(1):106-13. doi: 10.1016/j.otohns.2005.09.027. PMID 16399189
- [Background] Noordzij JP, Affleck BD. Coblation versus unipolar electrocautery tonsillectomy: a prospective, randomized, single-blind study in adult patients. Laryngoscope. 2006 Aug;116(8):1303-9. doi: 10.1097/01.mlg.0000225944.00189.e9. PMID 16885729
- [Background] Diakos EA, Gallos ID, El-Shunnar S, Clarke M, Kazi R, Mehanna H. Dexamethasone reduces pain, vomiting and overall complications following tonsillectomy in adults: a systematic review and meta-analysis of randomised controlled trials. Clin Otolaryngol. 2011 Dec;36(6):531-42. doi: 10.1111/j.1749-4486.2011.02373.x. PMID 21812940
- [Background] Thorneman G, Akervall J. Pain treatment after tonsillectomy: advantages of analgesics regularly given compared with analgesics on demand. Acta Otolaryngol. 2000 Oct;120(8):986-9. doi: 10.1080/00016480050218744. PMID 11200596
- [Background] Naesh O, Niles LA, Gilbert JG, Ammar MM, Phibbs PW, Phillips AM, Khrapov AV, Robert AJ, McClintock A. A randomized, placebo-controlled study of rofecoxib with paracetamol in early post-tonsillectomy pain in adults. Eur J Anaesthesiol. 2005 Oct;22(10):768-73. doi: 10.1017/s0265021505001274. PMID 16211736
- [Background] Hiller A, Silvanto M, Savolainen S, Tarkkila P. Propacetamol and diclofenac alone and in combination for analgesia after elective tonsillectomy. Acta Anaesthesiol Scand. 2004 Oct;48(9):1185-9. doi: 10.1111/j.1399-6576.2004.00473.x. PMID 15352967
- [Background] Salonen A, Kokki H, Nuutinen J. Recovery after tonsillectomy in adults: a three-week follow-up study. Laryngoscope. 2002 Jan;112(1):94-8. doi: 10.1097/00005537-200201000-00017. PMID 11802045
- [Background] Ashbach MN, Ostrower ST, Parikh SR. Tonsillectomy techniques and pain: a review of randomized controlled trials and call for standardization. ORL J Otorhinolaryngol Relat Spec. 2007;69(6):364-70. doi: 10.1159/000108369. Epub 2007 Nov 23. PMID 18033974